CLINICAL TRIAL: NCT01628367
Title: The Effectiveness of the Cytoplast Technique in Preventing Bone Loss Around Immediate Implant Placement in the Esthetic Zone. A Randomized Clinical Trial.
Brief Title: Guided Bone Regeneration Around Immediate Implants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Professor and Director of Graduate Periodontics, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00050746
Record Dates: First submitted 2012-06-11; First posted 2012-06-26 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-03-20 (Actual); Status verified 2017-02

CONDITIONS: Missing Tooth
MeSH Terms: conditions — Anodontia | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Membrane (Experimental): Test (membrane): Extraction and immediate implant placement will be performed. The gaps between the implant and socket walls will be filled with a bone graft material. Sites in the test group will receive a high-density PTFE (d-PTFE) membrane over the socket.
  Interventions: Procedure: Minimally Traumatic Tooth Extraction; Device: Immediate Implant Placement; Biological: Bone Graft Placement; Biological: Membrane placement; Drug: Medications
- Collagen plug (Active Comparator): Control (collagen plug): Extraction and immediate implant placement will be performed. The gaps between the implant and socket walls will be filled with a bone graft material. Sites in the control group will receive a collagen wound dressing over the socket.
  Interventions: Procedure: Minimally Traumatic Tooth Extraction; Device: Immediate Implant Placement; Biological: Bone Graft Placement; Biological: Collagen plug placement; Drug: Medications

INTERVENTIONS:
Procedure: Minimally Traumatic Tooth Extraction — The surgeon will perform a minimally traumatic tooth extraction in the following fashion. Intrasulcular incisions will be performed with at 15-C scalpel around the tooth to be extracted.
  A periotome will then be introduced into the periodontal ligament space in order to sever the subcrestal attachment and expand the periodontal ligament space. Elevators will be used to initiate luxation of teeth. After significant mobility has been achieved through elevation, forceps will be used only to deliver the tooth. Finally, the socket will be curetted to remove all granulomatous tissue and irrigated with sterile isotonic saline solution.
Device: Immediate Implant Placement — A threaded titanium alloy implant with an internal hex connection and a Resorbable Blast Texturing (RBT) surface (Tapered Internal® Implant System, Biohorizons, Inc., Birmingham, AL, USA) will be placed using a surgical guide. Implant diameter of 3.8mm with lengths of either 12 or 15mm will be used. Implants will be placed approximately 3-4mm below the free gingival margin or 2-3mm below the cemento-enamel junction of adjacent teeth.
Biological: Bone Graft Placement — Circumferential defects or dehiscences around the immediately placed implant will be grafted. enCore™ Combination Allograft (Osteogenics Biomedical, Lubbock, Texas, USA) will be used as the bone graft material.
Biological: Membrane placement — A non absorbable d-PTFE membrane (Cytoplast® TXT-200, Osteogenics Biomedical, Lubbock, Texas, USA) will be trimmed to an appropriate size and shape to completely cover the implant site, and extend about 3-5mm beyond on the facial aspect. The membrane will be tucked under the sub-periosteal flap. Care will be taken to ensure that the membrane is resting on bone all around the socket margins. The membrane will be kept a minimum of 1.5mm from the adjacent tooth roots in the interdental area.
  Arms: Membrane
Biological: Collagen plug placement — A bio-absorbable collagen wound dressing (CollaPlug®, Zimmer Dental, Carlsbad, CA, USA) will be trimmed to the appropriate size, so as to cover the socket
  Arms: Collagen plug
Drug: Medications — Patients will be given amoxicillin 500mg 2 days prior to the surgery and will then continue for every 8 hours for 10 days. Patients will also take Ibuprofen 600mg every 6 hours for the first 3 days following the surgery, and then as needed for pain. Patients will also receive a prescription for Vicodin as needed for pain, every 4 to 6 hours

SUMMARY:
An important result of healing after tooth extraction is a reduction in dimensions of the remaining bone at that site. This reduction of bone volume precludes successful restoration of the space using a dental implant. Bone augmentation has shown promise in clinical reports to reduce this loss of bone volume, thus allowing implant placement and restoration. The purpose of this study is to evaluate the clinical and radiographic outcomes of guided bone regeneration around dental implants placed in fresh extraction sockets.

DETAILED DESCRIPTION:
Aim: The purpose of this clinical study is to investigate the effect of a non-resorbable polytetrafluoroethylene (PTFE) membrane on immediate implant placement in the esthetic zone.

Material and Methods: Systemically healthy subjects presenting with a hopeless tooth in the maxillary premolar or anterior region will be recruited in the study. Following a minimally traumatic tooth extraction, subjects will be randomly distributed into one of two treatment groups, a Membrane (Test) or a No Membrane (Control) group. Both groups will receive immediate placement of an implant along with placement of a bone graft material to fill the spaces around the implant. Sites in the test group will receive a non-resorbable PTFE membrane over the socket, whereas those in the control group will receive a collagen dressing over the socket. At sites in the test group, the membrane will be removed at 4 weeks. A second stage surgery and placement of a provisional restoration will be carried out 4 months after implant placement. Final restorations will be placed 3 months after placement of the provisional restoration. Clinical and radiographic measurements will be performed at baseline, implant placement, placement of provisional and final restorations and at the 5-month recall visit.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 or older.
* Systemically healthy (American Society of Anesthesiologists I or II).
* Subjects will have one or more anterior or premolar teeth with a hopeless prognosis, with adjacent and opposing teeth present.
* Compliance with all requirements in the study and signing the informed consent

Exclusion Criteria:

* Active acute infection at the extraction site (e.g., sinus tract, swelling)
* Absence of sufficient mesio-distal width to place an implant as per the study protocol.
* Absence of sufficient bone height to house a 10mm long implant.
* The subject lacks a stable occlusion and/or a healthy periodontium.
* Current smokers or quit smoking less than one year
* Chronic use of medications known to affect the periodontal status (calcium antagonists, anticonvulsives, immunosuppressives, anti-inflammatory medications)
* Pregnancy or lactating mothers
* Current orthodontic or periodontal treatments
* History of alcoholism or drug abuse
* Untreated deep carious lesions or defective restorations that can potentially exacerbate during the course of the study
* Diseases of the immune system or any medical condition that may influence the outcome (uncontrolled diabetes (HbA1c >7)
* Bone disorders (hyperparathyroidism, osteoporosis, or Paget's disease)
* Neurologic or psychiatric disorders, systemic infections
* A history of IV bisphosphonate use.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS,MSD,PhD, Principal Investigator — Department of Periodontics and Oral Medicine, The University of Michigan, School of Dentistry
Locations (1):
- Graduate Periodontics Dept of Periodontics and Oral Medicine University of Michigan - School of Dentistry 1011 N. University, Room 1324, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Double-group, parallel, single-blinded, randomize clinical trial
Pre-assignment Details: Forty-eight patients were consented and screened; 35 initially included then 3 excluded based on socket morphology after extraction. Final enrollment = 32
Groups:
- Test: Membrane:
  Extraction and immediate implant placement will be performed. The gaps between the implant and socket walls will be filled with a bone graft material. Sites in the test group will receive a high-density PTFE (d-PTFE) membrane over the socket.
  Membrane placement: A non absorbable d-PTFE membrane (Cytoplast® TXT-200, Osteogenics Biomedical, Lubbock, Texas, USA) will be trimmed to an appropriate size and shape to completely cover the implant site, and extend about 3-5mm beyond on the facial aspect. The membrane will be tucked under the sub-periosteal flap. Care will be taken to ensure that the membrane is resting on bone all around the socket margins. The membrane will be kept a minimum of 1.5mm from the adjacent tooth roots in the interdental area.
- Control: Collagen plug:
  Extraction and immediate implant placement will be performed. The gaps between the implant and socket walls will be filled with a bone graft material. Sites in the control group will receive a collagen wound dressing over the socket.
  Collagen plug placement: A bio-absorbable collagen wound dressing (CollaPlug®, Zimmer Dental, Carlsbad, CA, USA) will be trimmed to the appropriate size, so as to cover the socket
Period: Overall Study
Arm/Group | Test | Control
Started | 16 | 16
Completed | 15 | 16
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test | Control | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Customized [Number; unit: participants]
  18 years old and older | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 14 | 12 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Mean keratanized gingiva (KG) width [Mean (Standard Deviation); unit: millimeters] — Width of the keratinized gingiva at one study site
  millimeters | 4.73 (1.83) | 3.63 (1.93) | 4.18 (1.88)
Soft tissue thickness [Mean (Standard Deviation); unit: millimeters]
  4mm from free gingival margin (FGM) | .97 (.23) | 1 (.18) | .985 (.59)
  6mm from free gingival margin (FGM) | 1.07 (.32) | 1.09 (.2) | 1.08 (.26)
Buccal plate thickness [Mean (Standard Deviation); unit: millimeters] — Thickness of the buccal plate measured clinically at the study site
  millimeters | .93 (.46) | .75 (.26) | .84 (.36)
Lingual plate thickness [Mean (Standard Deviation); unit: millimeters] — Thickness of the lingual plate measured clinically at the study site
  millimeters | 1.23 (.46) | .875 (.34) | 1.0525 (.4)
Teeth [Number; unit: Teeth] — Sites at which immediate implant were placed.
  Teeth
    Maxillary Anteriors | 5 | 5 | 10
    Maxillary Premolars | 9 | 5 | 14
    Mandibular Premolars | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Thickness of Buccal Bone
Description: Change of buccal bone volume over study duration
Time Frame: One year
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Test | Control
Number analyzed (Participants) | 15 | 16
millimeters
  4mm from free gingival margin (FGM) | .73 (.86) | .86 (.56)
  6mm from free gingival margin (FGM) | .63 (.75) | .66 (.77)

2. Secondary Outcome: Change in Interproximal Bone Levels
Description: Change of interproximal marginal bone loss (mean of mesial and distal sites)
Time Frame: One year
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Test | Control
Number analyzed (Participants) | 15 | 16
millimeters | 1.38 (.99) | 1.42 (.66)

3. Secondary Outcome: Pink Esthetic Score
Description: Pink esthetic score per Furhauser et.al. measured at study conclusion where based on seven variables: mesial papilla, distal papilla, soft-tissue level, soft-tissue contour, alveolar process deficiency, soft-tissue color and texture (Fig. 1). Each variable was assessed with a 2-1-0 score, with 2 being the best and 0 being the poorest score. Thus a maximum score of 14 is best, and 0 is the worst.
Time Frame: One year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Test | Control
Number analyzed (Participants) | 15 | 16
units on a scale | 11.53 (1.13) | 9.88 (2.13)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Test | Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (N=16) | Control (N=16)
Implant Failure (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No